CLINICAL TRIAL: NCT02559466
Title: Efficacy of Deep Transcranial Magnetic Stimulation (TMS) for Treatment-resistant Depression and Neuroanatomical Correlates: a Randomized Clinical Study Coupled With Positon Emission Tomography (PET)
Brief Title: Efficacy of Deep Transcranial Magnetic Stimulation (TMS) for Treatment-resistant Depression and Neuroanatomical Correlates: a Clinical Study Coupled With Positon Emission Tomography (PET)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-08; RCAPHM15_0084 (Other: APHM); 2015-A00345-44 (Registry Identifier: ID RCB)
Record Dates: First submitted 2015-09-23; First posted 2015-09-24 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Pharmacoresistant Depression
Keywords: pharmaco-resistant depressed patients
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients stimulated with a H-TMS (deep) (Experimental): 20 sessions navigated with Deep Transcranial Magnetic Stimulation
  Interventions: Device: Transcranial Magnetic Stimulation (TMS - ) - MagPro®; Device: Positon Emission Tomography (PET) - Discovery 710®
- Patients stimulated with a conventional TMS (Other): 20 sessions navigated with Conventional Transcranial Magnetic Stimulation
  Interventions: Device: Transcranial Magnetic Stimulation (TMS - ) - MagPro®; Device: Positon Emission Tomography (PET) - Discovery 710®

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation (TMS - ) - MagPro® — Class IIa
Device: Positon Emission Tomography (PET) - Discovery 710® — Class IB

SUMMARY:
Repetitive transcranial magnetic stimulation (TMS) is an emergent non-invasive treatment for treatment resistant depression (TRD). The exact neuro-functional mechanisms related to TMS efficiency remains however unknown; besides local effect on the target, TMS may induce interaction changes between remote cerebral regions. On the other hand, few studies have been performed in comparison to sham placebo stimulation. The investigators recently showed that non-responder depressive patients to TMS exhibited deeper and wider brain functional abnormalities hardly reachable by standard coils. The H1-Coil is a novel TMS (H-TMS) device capable of inducing a magnetic field with a deeper and wider distribution than standard coils.

The investigators design here a randomized controlled study in which the investigators will compare the clinical effects of H-coil TMS and standard TMS in patients with TRD, and their functional neuroanatomical correlates and changes in connectivity by Positron Emission Tomography (PET). The general objective is to better understand the mechanisms related to TMS efficiency in pharmacoresistant depression, in order to propose the best therapeutic approach for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients who met the diagnosis of major depressive episode (MDE)
* Patient right-handed
* Men and women aged over 18 years with major depressive episode IV (DSM-IV criteria), isolated or recurrent.
* Scores on the scale MADRS> 20
* Resistance Criterion defined as the failure of two antidepressants effective dose for a minimum of six weeks.
* Drug Therapy stable for at least 2 weeks

Exclusion Criteria:

* Bipolar disorder type I or type II
* Depression With Psychotic Features
* Diagnosis according comorbid Axis I (DSM IV) with schizophrenia, alcohol abuse and / or toxic substances.
* Inpatient under stress or under legal protection measure (guardianship, curatorship)
* Counter to the practice of Transcranial Magnetic Stimulation : a personal history of seizure, history of neurological or neurosurgical pathologies, metallic prosthetic material or foreign objects (pacemakers, prosthetic eye equipment, etc.).
* Pregnant or breastfeeding ongoing.
* Somatic disorder may affect cognitive abilities and brain structures
* Known allergy to any component of Fludeoxyglucose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-07-17 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
The depression score in Montgomery-Åsberg Depression Rating Scale (MADRS). | 24 month
  performed before and after TMS

SECONDARY OUTCOMES:
Short self-completion questionnaire on symptoms of depression | 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France